CLINICAL TRIAL: NCT01982058
Title: Intimacy-Enhancing Couples' Intervention for Localized Prostate Cancer
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Rutgers, The State University of New Jersey (Other)
Collaborators: Rutgers Cancer Institute of New Jersey (Other); Memorial Sloan Kettering Cancer Center (Other); Fox Chase Cancer Center (Other)
Responsible Party: Principal Investigator, Sharon Manne, PhD, Professor of Medicine, Rutgers, The State University of New Jersey
Allocation: Randomized | Model: Factorial | Masking: None | Purpose: Supportive Care
Other Study IDs: 0220100274; 0220100274 (Other: IRB number); NCI-2012-00552 (Other: CTRP (Clinical Trails Reporting Program)); 131023 (Other: Rutgers Cancer Institute of New Jersey)
Record Dates: First submitted 2013-06-24; First posted 2013-11-13 (Estimated); Last update posted 2022-10-19 (Actual); Status verified 2022-10

CONDITIONS: Prostate Cancer; Sexual Dysfunction and Infertility; Sexuality
MeSH Terms: conditions — Prostatic Neoplasms; Sexual Dysfunction, Physiological; Infertility; Sexuality | interventions — Counseling; Diet Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Intimacy-Enhancing Couples (Experimental): Patients and their partners receive communication and intimacy-enhancing intervention (IEC) once a week comprising the following five 90-minute sessions: Orientation and Stories of the Cancer Experience; Communication and Listening to Partner's concerns; Communication and Coping with Cancer Issues as a Team; Being Supportive to Solve Concerns; and Reflecting on Changes and Future Adaptation.
  Interventions: Other: communication intervention; Other: counseling intervention; Other: questionnaire administration
- General Health and Wellness (Active Comparator): Patients and their partners receive a General Health and Wellness intervention focusing on nutrition and physical activity once a week comprising of five 90-minute sessions: Introduction and Nutrition Basics; Nutrition and Prevention of Recurrence; Nutritional Review and Introduction to Relaxation; Physical Activity Basics; Aerobics and Resistance Exercises and Wrap up.
  Interventions: Other: counseling intervention; Other: nutrition intervention; Other: questionnaire administration
- Usual Care (Other): Patients and their partners receive standard psychological and emotional care (usual care [UC]) (i.e., social work consultations and referral to a psychiatrist or psychologist, if requested or deemed necessary by the attending physician).
  Interventions: Other: questionnaire administration

INTERVENTIONS:
Other: communication intervention
  Arms: Intimacy-Enhancing Couples
Other: counseling intervention
  Arms: General Health and Wellness; Intimacy-Enhancing Couples
Other: nutrition intervention
  Arms: General Health and Wellness
Other: questionnaire administration

SUMMARY:
RATIONALE: Participating in a therapy program may enhance communication and intimacy between men with prostate cancer and their partners.

PURPOSE: This randomized clinical trial is studying how well therapy enhances communication and intimacy for men with early stage prostate cancer and for their partners.

DETAILED DESCRIPTION:
Aim 1 A. To evaluate the impact of an Intimacy-Enhancing Couples' intervention (IEC) versus a General Health and Wellness Intervention (GHW) and a Usual care control (UC) on patient and partner psychological and relationship outcomes.

B. To determine whether relationship length, pre-intervention relationship satisfaction, and men's pre-intervention masculinity moderate the effects of IEC on couples' psychological and relationship outcomes

Aim 2 A. To evaluate whether IEC has an effect on couples' communication and intimacy when compared with GHW and UC and to determine whether changes in relationship communication and intimacy mediate changes in couples' psychological and relationship outcomes.

Exploratory Aim:

A. To evaluate the impact of IEC versus GHW on physical activity and fruit and vegetable intake as well as each partner's support for the other partner's adoption of greater physical activity and more fruit and vegetable intake.

ELIGIBILITY:
Inclusion Criteria:

* Patient has a primary diagnosis of localized prostate cancer (T1, T2, N=0 M=0, T3 N=0 M=0)
* Patient had surgery or initiated radiation treatment (brachytherapy or external beam radiation) or began pre-radiation Androgen deprivation therapy within the past 12 months.
* Patient is currently married or living with a partner, with relationship duration at least 1 year
* Patient and partner live within a 1 hour commuting distance to recruitment site
* Patient and partner read and speak English
* Patient has an Impact of Events Scale (IES) score greater than or equal to 16 and/or partner has an IES score greater than or equal to 17.

Exclusion Criteria:

* Patient had a previous definitive treatment for prostate cancer
* Patient has a concurrent diagnosis of another cancer (other than non-melanoma skin cancer)
* Partner is diagnosed with cancer (other than non-melanoma skin cancer)
* Patient or partner have a significant hearing impairment

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 483 (Actual)
Dates: Start 2011-08-18 (Actual); Primary Completion 2017-08-07 (Actual); Study Completion 2017-08-07 (Actual)

PRIMARY OUTCOMES:
Psychological Functioning | 5 years
  General psychological functioning is assessed by the MHI-38 and the PHQ-9. Cancer-Specific distress is assessed by using the Impact of Events Scale Revised Cancer-Specific concerns is assessed with a 10 item assessment of commonly-experienced problems.
Relationship Functioning | 5 years
  Relationship satisfaction is assessed using the Dyadic Adjustment Scale

SECONDARY OUTCOMES:
Intimacy | 5 years
  General Relationship Intimacy. The Personal Assessment of Intimacy in Relationships Intimacy scale (PAIR) (94) is a 6 item scale assessing emotional closeness. Cancer-specific Relationship Intimacy (95-96) Participants rate the degree to which they felt close to and emotionally intimate with their partner during discussions about the cancer experience.
Relationship Communication | 5 years
  Perceived self-disclosure. The scale assesses the degree to which they disclose thoughts, information, and feelings about the cancer experience in the past week.
  Perceived partner disclosure. The scale assesses the degree to which their partner disclosed thoughts, information, and feelings.
  Perceived partner responsiveness. The scale assesses the degree to which the participant felt their partner understood and empathized with their disclosures.Mutual Constructive Communication. This subscale of the Communication Pattern Questionnaire (CPQ) is a 5-item scale that has been adapted.
  Holding back. Participants rate the degree to which they held back from talking to their partner about 11 domains of concern.
  Demand-Withdraw. The CPQ Demand-Withdraw subscale is a 6-item scale adapted.
  Mutual Avoidance. The CPQ Mutual Avoidance subscale is an adapted 6-item scale.

CONTACTS AND LOCATIONS:
Overall Officials: Sharon L Manne, Ph.D., Principal Investigator — Rutgers Cancer Institute of New Jersey
Locations (6):
- United States (6):
  - Rutgers Cancer Institute of New Jersey, New Brunswick, New Jersey
  - The University Hospital, Newark, New Jersey
  - Garden State Urology, Whippany, New Jersey
  - Memorial Sloan-Kettering Cancer Center, New York, New York
  - Hospital of the University of Pennsylvania, Philadelphia, Pennsylvania
  - Fox Chase Cancer Center, Philadelphia, Pennsylvania

IPD SHARING:
Plan to Share IPD: No